CLINICAL TRIAL: NCT02008877
Title: A Phase I/II Trial of Ganetespib in Combination With the mTOR Inhibitor Sirolimus for Patients With Recurrent or Refractory Sarcomas Including Unresectable or Metastatic Malignant Peripheral Nerve Sheath Tumors
Brief Title: SARC023: Ganetespib and Sirolimus in Patients With MPNST (Malignant Peripheral Nerve Sheath Tumors)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Collaborators: Synta Pharmaceuticals Corp. (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARC023; CDMRP-NF120087 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2013-11-25; First posted 2013-12-11 (Estimated); Results first posted 2019-05-02 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-04

CONDITIONS: Malignant Peripheral Nerve Sheath Tumors (MPNST); Sarcoma
Keywords: Malignant Peripheral Nerve Sheath Tumors; MPNST; Sarcoma; Ganetespib; Sirolimus; mTOR inhibitor; Heat shock protein; Hsp90
MeSH Terms: conditions — Neurofibrosarcoma; Sarcoma | interventions — STA 9090; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ganetespib / sirolimus (Experimental): 28-day cycles of ganetespib + sirolimus
  Interventions: Drug: ganetespib; Drug: Sirolimus

INTERVENTIONS:
Drug: ganetespib — Phase 1 Dose 1: 150 mg/m² IV on days 1, 8, and 15 intravenously over 1 hour; Phase 1 Dose 2: 200 mg/m² IV on days 1, 8, and 15 intravenously over 1 hour; Phase 2: 200 mg/m² IV on days 1, 8, and 15 intravenously over 1 hour
  Other Names: STA-9090
Drug: Sirolimus — 4mg taken orally once daily on a continuous dosing schedule; Loading dose 12 mg on cycle 1 day 1 only.
  Other Names: Rapamycin

SUMMARY:
Phase 1: To assess the safety, tolerability, and maximum tolerated dose (MTD)/ recommended dose of ganetespib when administered in combination with sirolimus in patients with refractory or relapsed sarcomas including unresectable or metastatic sporadic or neurofibromatosis type 1 (NF1) associated MPNST. Phase I enrollment has been closed.

Phase 2: To determine the clinical benefit of ganetespib in combination with sirolimus for patients with unresectable or metastatic sporadic or NF1 associated MPNST.

DETAILED DESCRIPTION:
Previously, no targeted agents have been able to cause tumor regression in a genetically engineered MPNST mouse model or human MPNST. Recently published data from Dr. Cichowski's laboratory demonstrated using Hsp90 inhibitors to enhance endoplasmic reticulum stress coupled with the mammalian target of rapamycin (mTOR) inhibitor sirolimus led to dramatic tumor shrinkage in a transgenic MPNST mouse model, which correlated with profound damage to the endoplasmic reticulum and cell death. Ganetespib is a novel, injectable, small molecule inhibitor of Hsp90 and is currently being investigated in adults with a broad range of tumor types with a favorable safety profile and promising early results. Ganetespib has been studied in preclinical in vivo models with a variety of targeted agents with no marked apparent pharmacological interactions. Sirolimus is a commercially available orally administered mTOR inhibitor and is the active metabolite of temsirolimus, which is FDA approved agent for advanced metastatic renal cell carcinoma. Sirolimus has been studied and tolerated in combination with multiple cytotoxic and targeted agents in a variety of tumor types. Based on strong preclinical rationale, the investigators hypothesize that ganetespib in combination with sirolimus will cause tumor regression in patients with refractory MPNSTs.

The investigators propose a multi-institutional open label phase I/II trial of ganetespib in combination with sirolimus in patients with refractory sarcoma including MPNST. Hsp90 inhibitors and mTOR inhibitors have also both demonstrated benefit in a variety of preclinical bone and soft tissue sarcoma models. The investigators hypothesize that these agents that work on separate and potentially synergistic pathways will also be beneficial for other refractory bone and soft tissue sarcomas. Thus, the phase I component will be open to patients with refractory sarcomas, which will also expedite enrollment. Upon determination of the recommended dosing, a phase II study will be conducted. The phase II study population will be limited to patients with a diagnosis of MPNST.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 16 years old
* Patients with unresectable or metastatic histologically confirmed sporadic or NF1 associated high grade MPNST
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Patients must have at least 1 measurable tumor
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy (toxicity < grade 2)
* Must be able to swallow whole pills
* Adequate organ function
* Normal fasting cholesterol and triglycerides
* May be on cholesterol medications

Exclusion Criteria:

* Patients receiving current treatment with corticosteroids or another immunosuppressive. Topical or inhaled corticosteroids are allowed.
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Symptomatic congestive heart failure
* Severely impaired lung function
* Significant vascular disease
* Uncontrolled diabetes
* Active (acute or chronic) or uncontrolled severe infections hepatitis
* Impairment of gastrointestinal function
* Patients with an active, bleeding diathesis or significant coagulopathy
* Use of cytochrome P450 isoenzyme 3A4 (CYP3A4)/ CYP2C19 substrates

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12; Primary Completion 2018-04 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AeRang Kim, MD, PhD, Principal Investigator — Children's National Research Institute; Brigitte Widemann, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (7):
- United States (7):
  - Sarcoma Oncology Center, Santa Monica, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Iowa, Iowa City, Iowa
  - National Cancer Institute, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- [Derived] Kim A, Lu Y, Okuno SH, Reinke D, Maertens O, Perentesis J, Basu M, Wolters PL, De Raedt T, Chawla S, Chugh R, Van Tine BA, O'Sullivan G, Chen A, Cichowski K, Widemann BC. Targeting Refractory Sarcomas and Malignant Peripheral Nerve Sheath Tumors in a Phase I/II Study of Sirolimus in Combination with Ganetespib (SARC023). Sarcoma. 2020 Jan 30;2020:5784876. doi: 10.1155/2020/5784876. eCollection 2020. PMID 32089640
- See also: SARC Website — http://www.sarctrials.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Dose 1: For each 28-day cycle, subjects took doses of both ganetespib + sirolimus:
  ganetespib: 150 mg/m² IV on days 1, 8, and 15 intravenously over 1 hour
  Sirolimus: 4mg taken orally once daily on a continuous dosing schedule; Loading dose 12 mg on cycle 1 day 1 only.
- Phase 1 Dose 2; Phase 2: For each 28-day cycle, subjects took doses of both ganetespib + sirolimus:
  ganetespib: 200 mg/m² IV on days 1, 8, and 15 intravenously over 1 hour
  Sirolimus: 4mg taken orally once daily on a continuous dosing schedule; Loading dose 12 mg on cycle 1 day 1 only.
Period: Overall Study
Arm/Group | Phase 1 Dose 1 | Phase 1 Dose 2 | Phase 2
Started | 3 | 7 | 10
Completed | 3 | 6 | 10
Not Completed | 0 | 1 | 0
Not completed — Inevaluable | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ganetespib / Sirolimus: 28-day cycles of ganetespib + sirolimus
  ganetespib: 200 mg/m² IV on days 1, 8, and 15 intravenously over 1 hour
  Sirolimus: 2mg taken orally once daily on a continuous dosing schedule; Loading dose 12 mg on cycle 1 day 1 only.
Arm/Group | Ganetespib / Sirolimus
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] — Population: 10 patients were enrolled in Phase 1 and 10 patients were enrolled in Phase 2 of the study. Overall number of patients enrolled was 20.
  years
    Phase I: number analyzed (Participants) | 10
    Phase I | 26 [16 to 89]
    Phase 2: number analyzed (Participants) | 10
    Phase 2 | 38 [24 to 61]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 10 patients were enrolled in Phase 1 and 10 patients were enrolled in Phase 2 of the study. Overall number of patients enrolled was 20.
  Participants
    Phase I: number analyzed (Participants) | 10
    Phase I: Female | 2
    Phase I: Male | 8
    Phase 2: number analyzed (Participants) | 10
    Phase 2: Female | 4
    Phase 2: Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 0
  Unknown or Not Reported | 2
Sarcoma subtype [Count of Participants; unit: Participants] — Population: 10 patients were enrolled in Phase 1 and 10 patients were enrolled in Phase 2 of the study. Overall number of patients enrolled was 20.
  Participants
    Phase I: number analyzed (Participants) | 10
    Phase I: Alveolar soft part sarcoma | 1
    Phase I: Ewing sarcoma | 1
    Phase I: Leiomyosarcoma | 2
    Phase I: Liposarcoma | 3
    Phase I: MPNST NF1 Associated | 3
    Phase I: MPNST Sporadic | 0
    Phase 2: number analyzed (Participants) | 10
    Phase 2: Alveolar soft part sarcoma | 0
    Phase 2: Ewing sarcoma | 0
    Phase 2: Leiomyosarcoma | 0
    Phase 2: Liposarcoma | 0
    Phase 2: MPNST NF1 Associated | 5
    Phase 2: MPNST Sporadic | 5
Tumor location at diagnosis [Count of Participants; unit: Participants] — Population: 10 patients were enrolled in Phase 1 and 10 patients were enrolled in Phase 2 of the study. Overall number of patients enrolled was 20.
  Participants
    Phase I: number analyzed (Participants) | 10
    Phase I: Abdomen | 1
    Phase I: Extremity | 1
    Phase I: Head | 1
    Phase I: Lung | 0
    Phase I: Mediastinum | 1
    Phase I: Peritoneum | 1
    Phase I: Skin | 1
    Phase I: Spine | 1
    Phase I: Other | 3
    Phase 2: number analyzed (Participants) | 10
    Phase 2: Abdomen | 1
    Phase 2: Extremity | 4
    Phase 2: Head | 0
    Phase 2: Lung | 1
    Phase 2: Mediastinum | 0
    Phase 2: Peritoneum | 0
    Phase 2: Skin | 0
    Phase 2: Spine | 2
    Phase 2: Other | 2
History of metastatic disease [Count of Participants; unit: Participants] — Population: 10 patients were enrolled in Phase 1 and 10 patients were enrolled in Phase 2 of the study. Overall number of patients enrolled was 20.
  Participants
    Phase 1: number analyzed (Participants) | 10
    Phase 1 | 9
    Phase 2: number analyzed (Participants) | 10
    Phase 2 | 9
Prior chemotherapy regimen [Count of Participants; unit: Participants] — Population: 10 patients were enrolled in Phase 1 and 10 patients were enrolled in Phase 2 of the study. Overall number of patients enrolled was 20.
  Participants
    Phase 1: number analyzed (Participants) | 10
    Phase 1 | 10
    Phase 2: number analyzed (Participants) | 10
    Phase 2 | 8
Prior radiation [Count of Participants; unit: Participants] — Population: 10 patients were enrolled in Phase 1 and 10 patients were enrolled in Phase 2 of the study. Overall number of patients enrolled was 20.
  Participants
    Phase 1: number analyzed (Participants) | 10
    Phase 1 | 7
    Phase 2: number analyzed (Participants) | 10
    Phase 2 | 6
Prior surgery [Count of Participants; unit: Participants] — Population: 10 patients were enrolled in Phase 1 and 10 patients were enrolled in Phase 2 of the study. Overall number of patients enrolled was 20.
  Participants
    Phase 1: number analyzed (Participants) | 10
    Phase 1 | 10
    Phase 2: number analyzed (Participants) | 10
    Phase 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicities of Ganetespib When Administered in Combination With Sirolimus.
Description: To assess the safety, tolerability, and maximum tolerated/ recommended dose of ganetespib when administered in combination with sirolimus in patients with refractory sarcomas or unresectable or metastatic sporadic or neurofibromatosis type 1 (NF1) associated MPNST. Toxicities observed during the first cycle will be used to define the MTD/Recommended dose. Toxicity will be graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. DLT will be defined as any of the following events that are possibly, probably, or definitely attributable to ganetespib or sirolimus. The DLT observation period for the purposes of dose escalation will be the first cycle of therapy.
Time Frame: Toxicities will be evaluated over the first treatment cycle (each cycle=28 days)
Population: 10 patients were enrolled in Phase 1 of the study to determine MTD/RD. Three patients were enrolled in the first dose level. Six patients were enrolled at dose level 2. 1 patient was inevaluable.
Measure: Number; unit: DLTs
Arm/Group | Ganetespib / Sirolimus
Number analyzed (Participants) | 9
DLTs
  Dose Level 1: number analyzed (Participants) | 3
  Dose Level 1 | 0
  Dose Level 2: number analyzed (Participants) | 6
  Dose Level 2 | 1

2. Primary Outcome: Clinical Benefit of Ganetespib in Combination With Sirolimus
Description: Assessed using the World Health Organization (WHO) criteria. Tumor assessments will be obtained every 2 cycles. Clinical benefit is defined as stable disease, Partial Response (PR), Complete Response (CR). For patients who experience progression by WHO but in the opinion of the treating investigator are deriving benefit from therapy and have not otherwise met off treatment or off study criteria, may continue on treatment as long as patient has not met progression by RECIST 1.1.
Time Frame: Response evaluations will be performed after every 2 treatment cycles (each cycle=28 days)
Population: 10 patients were enrolled in Phase 1 and 10 patients were enrolled in Phase 2 of the study. Overall number of patients enrolled was 20.
Measure: Count of Participants; unit: Participants
Arm/Group | Ganetespib / Sirolimus
Number analyzed (Participants) | 20
Participants
  Phase 1: number analyzed (Participants) | 10
  Phase 1 | 1
  Phase 2: number analyzed (Participants) | 10
  Phase 2 | 0

3. Secondary Outcome: Change in Plasma Pharmacokinetic Profile of Ganetespib and Sirolimus When Administered in Combination-Observed Maximum Plasma Concentration (Cmax)
Description: To describe the plasma pharmacokinetic profile of ganetespib and sirolimus when administered in combination therapy.
Time Frame: Pre-therapy levels drawn at baseline and pharmacokinetic analysis occurs on Cycle 1 Day 15
Population: 10 patients were enrolled in Phase 1 of the study. Three patients were enrolled in the first dose level. Six patients were enrolled at dose level 2. 1 patient was inevaluable.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ganetespib / Sirolimus
Number analyzed (Participants) | 9
ng/mL
  Dose Level 1- Sirolimus trough: number analyzed (Participants) | 3
  Dose Level 1- Sirolimus trough | 12.1 (3.6)
  Dose Level 2- Sirolimus trough: number analyzed (Participants) | 6
  Dose Level 2- Sirolimus trough | 12.5 (8.9)

4. Secondary Outcome: Changes in Pharmacodynamic Parameters in Peripheral Blood Mononuclear Cells
Description: To explore changes in pharmacodynamic parameters in peripheral blood mononuclear cells performed on day 1 prior to ganetespib and sirolimus administration, and on day 15, 6 hours post drug administration. Hsp inhibition (Hsp70), mTOR inhibition (phospho-S6 and Akt Phosphorylation), UPR activation (EIF2alpha phosphorylation) will be explored. Western blot analyses were performed for phospho (p)-Akt, p-eIF2α, p-S6, and Hsp70. The absorbance of each phosphoprotein lane was recorded and protein levels were determined after normalizing for levels of corresponding total protein.
Time Frame: Baseline and Cycle 1 Day 15
Population: 11 subjects provided consent and had adequate specimens for analysis.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Ganetespib / Sirolimus
Number analyzed (Participants) | 11
ratio
  Hsp70 at Baseline | 0.81 (0.39)
  Hsp70 at Cycle 1 Day 15 | 0.84 (0.56)
  pAKT at Baseline | 1.20 (0.70)
  pAKT at Cycle 1 Day 15 | 1.44 (1.00)
  p-S6 at Baseline | 1.25 (0.40)
  p-S6 at Cycle 1 Day 15 | 0.54 (0.24)
  p-eiF2alpha at Baseline | 1.02 (0.26)
  p-eiF2alpha at Cycle 1 Day 15 | 0.49 (0.22)

5. Secondary Outcome: Patient-reported Pain Severity and the Impact of Pain on Daily Activities
Description: To assess patient-reported pain severity and the impact of pain on daily activities before and during treatment with ganetespib and sirolimus. The Numerical Rating Scale-11 (NRS-11) will be used to assess pain severity. The NRS-11 is a self-report segmented 11-point numeric scale that assesses pain severity. It consists of a horizontal line with 0 representing "no pain" at the right end of the line and 10 representing "worst pain you can imagine" at the left end.The Brief Pain Inventory is a 7-item self-report questionnaire that measures the extent to which pain interferes with daily functioning. Patients are asked to indicate how much pain interfered with various activities in the past week, with scores ranging from 0 (does not interfere) to 10 (completely interferes). A total score is obtained by taking the mean of the scores for all 7 items; thus, the total pain interference score can range from 0 to 10.
Time Frame: Baseline and prior to Cycle 3
Population: Thirteen subjects in phase 1 and phase 2 cohorts combined had MPNST and completed the pain evaluations. 4/13 subjects completed both baseline and pre-cycle 3 evaluations for pain.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ganetespib / Sirolimus
Number analyzed (Participants) | 4
units on a scale
  Baseline- Overall pain intensity | 7.5 [0 to 10]
  Baseline- Tumor pain intensity | 7.5 [0 to 10]
  Baseline- Pain interference | 6.49 [0 to 10]
  Prior to Cycle 3- Overall pain intensity | 5 [0 to 10]
  Prior to Cycle 3- Tumor pain intensity | 4.75 [0 to 10]
  Prior to Cycle 3- Pain interference | 3.14 [0 to 10]

6. Secondary Outcome: Utility of Three-dimensional MRI (3D-MRI) Analysis in Comparison to 1-dimensional and 2-dimensional Measurements
Description: To evaluate the utility of three-dimensional MRI (3D-MRI) analysis in comparison to 1-dimensional and 2-dimensional measurements as a method to more sensitively monitor response.
Time Frame: 4 months
Population: The 3D-MRI were not measurable with current modalities. Due to their nature and incomplete imaging, volumetric analysis was not feasible.
Arm/Group | Ganetespib / Sirolimus
Number analyzed (Participants) | 0

7. Secondary Outcome: Plasma Pharmacokinetic Profile of Ganetespib When Administered in Combination With Sirolimus
Description: To describe the plasma pharmacokinetic profile of ganetespib in terms of half life.
Time Frame: Cycle 1 Day 15
Population: 10 patients were enrolled in Phase 1 of the study. 1 patient was inevaluable.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ganetespib / Sirolimus
Number analyzed (Participants) | 9
hours
  Ganetespib half life for dose level 1: number analyzed (Participants) | 3
  Ganetespib half life for dose level 1 | 6.4 (2.1)
  Ganetespib half life for dose level 2: number analyzed (Participants) | 6
  Ganetespib half life for dose level 2 | 6.0 (0.9)

8. Secondary Outcome: Determine Maximum Tolerated Dose (MTD)/Recommended Dose (RD) of Ganetespib
Description: A conventional 3+3 dose escalation design was used for phase 1. All patients in phase 2 were treated with the recommended dose.
Time Frame: Phase 1 of study
Population: 1 patient was inevaluable in Phase 1 of study. The recommended dose of ganetespib was determined to be 200 mg/m2 intravenously on days 1, 8, 15 with sirolimus 4mg orally once daily with a cycle 1 day 1 loading dose of 12mg. All patients in phase 2 were treated with the recommended dose.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 Dose Level 1: For each 28-day cycle, subjects took doses of both ganetespib + sirolimus:
  ganetespib: 150 mg/m² IV on days 1, 8, and 15 intravenously over 1 hour
  Sirolimus: 4mg taken orally once daily on a continuous dosing schedule; Loading dose 12 mg on cycle 1 day 1 only.
- Phase 1 Dose Level 2; Phase 2: For each 28-day cycle, subjects took doses of both ganetespib + sirolimus:
  ganetespib: 200 mg/m² IV on days 1, 8, and 15 intravenously over 1 hour
  Sirolimus: 4mg taken orally once daily on a continuous dosing schedule; Loading dose 12 mg on cycle 1 day 1 only.
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 2
Number analyzed (Participants) | 3 | 6 | 10
Participants | 3 | 6 | 10

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Phase 1 Dose 1 | Phase 1 Dose 2 | Phase 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/7 | 1/10
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/7 | 6/10
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose 1 (N=3) | Phase 1 Dose 2 (N=7) | Phase 2 (N=10)
Gastrointestinal disorders- other (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate Aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gastric obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose 1 (N=3) | Phase 1 Dose 2 (N=7) | Phase 2 (N=10)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 (0) | 2 (2) | 3 (3)
Alanine Aminotransferase increased (Investigations) | 1 (3) | 1 (2) | 2 (8)
Alkaline Phosphatase increased (Investigations) | 1 (1) | 1 (2) | 5 (9)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (4) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Aspartate Aminotransferase increased (Investigations) | 2 (2) | 1 (2) | 3 (6)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (2)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
High cholesterol (Investigations) | 0 (0) | 2 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
CPK increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (5) | 7 (11) | 8 (14)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 2 (3) | 1 (1)
Edema trunk (General disorders) | 0 (0) | 1 (1) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (3) | 1 (1) | 6 (6)
Fever (General disorders) | 0 (0) | 1 (1) | 2 (2)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders-other (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
General disorders and admin site conditions-other (General disorders) | 1 (3) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 2 (4) | 3 (3) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3) | 2 (3) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (4)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Infections and infestations-other (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Investigations-other (Investigations) | 1 (1) | 0 (0) | 0 (0)
Irritability (General disorders) | 0 (0) | 1 (2) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (3) | 3 (8) | 4 (8)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 2 (4) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder-other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 3 (3) | 7 (9)
Neutrophil count decreased (Investigations) | 1 (3) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 3 (7) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Respiratory, thoracic and mediastinal disorders-other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Skin and subcutaneous tissue disorders-other (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Surgical and medical procedures-other (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 5 (6)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 2 (3) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-13): https://cdn.clinicaltrials.gov/large-docs/77/NCT02008877/Prot_SAP_000.pdf